CLINICAL TRIAL: NCT04971161
Title: A Randomized, Placebo-Controlled, Double-blind, Dose-Ranging, Multicenter, Phase IIb Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-CVU on Wound Healing of Therapy-Resistant Chronic Venous Ulcer (CVU)
Brief Title: Allogeneic ABCB5-positive Dermal Mesenchymal Stromal Cells for Treatment of CVU (Phase IIb)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: allo-APZ2-CVU-IIb; 2023-510162-27-00 (EU CTIS Number); U1111-1301-6596 (Registry Identifier: World Health Organization [WHO] Registry Network); 2020-004960-24 (EudraCT Number)
Record Dates: First submitted 2021-06-07; First posted 2021-07-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Skin Ulcer Venous Stasis Chronic
Keywords: Chronic Venous Ulcer; ABCB5; Allogeneic; Dermal mesenchymal stromal cells; varicose ulcer; skin ulcer; advanced therapy medicinal product; somatic cell therapy; phase IIb
MeSH Terms: conditions — Varicose Ulcer; Skin Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, dose-ranging, interventional, multicenter, phase IIb clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- allo-APZ2-CVU (dose group 1: 1 x 10e6 cells/cm²) (Experimental): Application of IMP on patients wound
  Interventions: Biological: allo-APZ2-CVU
- Placebo (Placebo Comparator): Application of IMP on patients wound
  Interventions: Drug: Placebo
- allo-APZ2-CVU (dose group 2: 3 x 10e6 cells/cm²) (Experimental): Application of IMP on patients wound
  Interventions: Biological: allo-APZ2-CVU
- allo-APZ2-CVU (dose group 3: 6 x 10e6 cells/cm²) (Experimental): Application of IMP on patients wound
  Interventions: Biological: allo-APZ2-CVU

INTERVENTIONS:
Biological: allo-APZ2-CVU — Suspension of ABCB5-positive dermal mesenchymal stromal cells. One topical application with a syringe.
  Other Names: Skin-derived ABCB5-positive dermal mesenchymal stromal cells
  Arms: allo-APZ2-CVU (dose group 1: 1 x 10e6 cells/cm²); allo-APZ2-CVU (dose group 2: 3 x 10e6 cells/cm²); allo-APZ2-CVU (dose group 3: 6 x 10e6 cells/cm²)
Drug: Placebo — One topical application with a syringe
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring the wound size reduction of CVUs) and safety (by monitoring adverse events [AEs]) of three dose groups of the investigational medicinal product (IMP) allo-APZ2-CVU, topically administered on target wounds of patients with CVU compared to placebo.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, dose-ranging, multicenter, phase IIb clinical trial to investigate the efficacy and safety of the IMP allo-APZ2-CVU on wound healing in patients with therapy-resistant CVU. The allogeneic IMP allo-APZ2-CVU contains skin-derived ABCB5-positive dermal mesenchymal stromal cells isolated from skin tissue of healthy donors and stored in a donor cell bank.

Patients will be randomized to be treated with allo-APZ2-CVU (dose 1, dose 2, dose 3) or placebo (50 patients per dose group). The patients will undergo treatment with the IMP on Day 0 (V3) and will be followed up for efficacy for 18 weeks (V4 until V14). Two safety follow-up visits will be performed at Month 6 (V15) and Month 10 (V16). An additional visit (V17) will be performed to follow up on target wounds of all patients who reached the primary endpoint (i.e. wound was closed at V13 and V14) at Month 16 (at least).

The wound healing process will be documented by standardized photography. The wound size measurement will start at the first Screening Visit (V1) and will be measured at each following on-site visit.

Pain will be assessed using a numerical rating scale and quality of life will be investigated with standardized and validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years old;
2. Chronic venous leg ulcer (as defined by the current AWMF guidelines: therapy-resistant ulcer that shows no tendency to heal within 3 months despite of optimal phlebological therapies or has not fully healed within 12 months) at lower leg and/or ankle region and has not been present longer than 15 years, diagnosed by doppler or duplex sonography, ankle brachial index (ABI, 0.9-1.3), physical examination and dermatological review;
3. Wound size of target ulcer between 1 and 50 cm² measured by a standardized photography at the screening visit;
4. If patients have 2 or more ulcers at the same extremity, the target ulcer has to be separated by a minimum bridge of 1 cm of epithelialized skin from other ulcers (the largest ulcer should be the target ulcer, if not decided otherwise at discretion of the investigator; the target ulcer is defined at Visit 1);
5. Body mass index between 15 and 50 kg/m²;
6. Patients understand the nature of the procedure and are providing written informed consent prior to any clinical trial procedure;
7. Women of childbearing potential must have a negative blood pregnancy test at Visit 1;
8. Women of childbearing potential and their partner must be willing to use highly effective contraceptive methods during the course of the clinical trial.

Exclusion Criteria:

1. Evidence of the ulcer extending to the underlying muscle, tendon, or bone;
2. Diabetes mellitus that has to be confirmed by blood test (Hemoglobin A1c >7.5%);
3. Peripheral Artery Disease including claudication with need of treatment;
4. Acute deep vein thrombosis (maximum 30 days from diagnosis) or a still untreated deep vein thrombosis;
5. Unable to tolerate leg ulcer compression bandage;
6. Infection of the target ulcer requiring treatment as judged clinically;
7. All diagnosed disorders, unrelated to CVU, that are influencing wound healing of the target wound at investigator's discretion;
8. Current use of medications that influence wound healing: systemic immunosuppressives, cytotoxic medicinal products, and systemic steroids (above Cushing-threshold level);
9. Patient who, in the opinion of the investigator, for any reason are unable or unwilling to complete the trial per protocol (e.g. alcohol or substance abuse, not mobile, short life expectancy) or there is evidence of any other medical condition (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
10. Any malignancy within the past 5 years, excluding successfully treated carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin without evidence of metastases;
11. Pregnant or lactating women;
12. Any known allergies to components of the IMP;
13. Prior surgical procedures such as bypass or mesh-graft treatment at target leg within 2 months prior to Visit 1 at target leg;
14. Patients with significant ulcer healing or wound size enlargement of more than 25% at Visit 2 compared to Visit 1;
15. Treatment of target ulcer with active wound care agents (e.g. Iruxol®N), which have not been paused 14 days before IMP application;
16. Current or previous (within 30 days of enrollment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
17. Previous participation in this clinical trial (except for screening failures due to an inclusion or exclusion criterion);
18. Employees of the sponsor, or employees or relatives of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Complete wound closure at Week 18 already persisting for at least two weeks | Week 18
  Complete wound closure at Week 18 already persisting for at least two weeks will be evaluated.
Assessment of adverse event (AE) occurrence | Up to 10 months
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Wound size change in percent at each post-baseline follow-up visit | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10
  Wound size change in percent at each post-baseline follow-up visit will be evaluated.
Time to complete wound closure | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10
  Time to complete wound closure will be evaluated.
Complete wound closures at each post-baseline follow-up visit | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10, Month 16
  Complete wound closures at each post-baseline follow-up visit will be evaluated.
Duration of wound closure | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10
  Duration of wound closure will be evaluated.
Recurrence of the wound | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10, Month 16
  Recurrence of the wound will be evaluated.
Quality of wound healing (wound exudate) at each post-baseline follow-up visit | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10, Month 16
  The Quality of wound healing will be assessed at each post-baseline follow-up visit on the basis of the amount and type of wound exudate.
Quality of wound healing (granulation tissue together with epithelialization) at each post-baseline follow-up visit | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10
  The Quality of wound healing will be assessed at each post-baseline follow-up visit on the basis of the formation of granulation tissue together with epithelialization.
Quality of wound healing (scar formation) at each post-baseline follow-up visit | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10
  The Quality of wound healing will be assessed at each post-baseline follow-up visit on the basis of the questions regarding scar formation.
Assessment of Quality of Life using the Wound-Quality of Life Questionnaire at V8, V11, V14, V15, V16 | Week 6, 12, 18, Month 6 and 10
  Quality of Life using the Wound-Quality of Life Questionnaire at V8, V11, V14, V15, V16 will be evaluated.
Pain assessment as per numerical rating scale on each post-baseline follow-up visit | Day 1-2, Week 1, 2, 4, 6, 8, 10, 12, 14, 16, Month 6 and 10
  Pain assessment as per numerical rating scale on each post-baseline follow-up visit will be evaluated.
Physical examination and vital signs at V14 | Week 18
  A physical body examination (e.g. general appearance, thyroid, head, lungs and thorax, ears, cardiovascular system, eyes, abdomen, nose-mouth-throat, musculoskeletal system, skin, extremities, lymph nodes, neurological system) will be performed and abnormal physical examination results will be evaluated and reported as AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kerstan, Dr., Principal Investigator — Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Würzburg
Locations (38):
- Germany (38):
  - MVZ Gefäßzentrum Aachen am Marienhospital Aachen GmbH, Aachen
  - Universitätsklinikum Augsburg, Klinik für Dermatologie und Allergologie, Campus Süd, Augsburg
  - Fachklinik Bad Bentheim, Dermatologische Ambulanz, Bad Bentheim
  - Helios Klinikum Berlin-Buch, Klinik für Plastische und Ästhetische Chirurgie, Berlin
  - Helios Klinikum Emil von Behring, Klinik für Plastische und Ästhetische Chirurgie, Berlin
  - Hautarztpraxis Dr. Niesmann & Dr. Othlinghaus, Hautzentrum im Jahrhunderthaus, Bochum
  - Katholisches Klinikum Bochum gGmbH, Venenzentrum der Kliniken für Dermatologie und Gefäßchirurgie der Ruhr-Universität Bochum, Bochum
  - Hautärzte Braunschweig am Altstadtmarkt, Hautärztliche Gemeinschaftspraxis, Braunschweig
  - Klinikum Bremerhaven Reinkenheide gGmbH, Klinik für Dermatologie, Allergologie und Phlebologie, Wundzentrum, Bremerhaven
  - Klinische Forschung Dresden GmbH, Dresden
  - Universitätsklinikum Erlangen, Hautklinik - Wundzentrum Dermatologie, Erlangen
  - Universitätsklinikum Essen, Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Essen
  - Universitätsklinikum Freiburg, Klinik für Dermatologie und Venerologie, Freiburg im Breisgau
  - Marienhospital Gelsenkirchen GmbH, Klinik für Chirurgie (Allgemein-, Viszeral- und Endokrine Chirurgie, Thorax-, Gefäß- und Endovaskuläre Chirurgie und Kinderchirurgie), Gelsenkirchen
  - SRH Wald-Klinikum Gera GmbH, Zentrum für Klinische Studien, Gera
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Hautkrankheiten, Greifswald
  - Praxis Dr. med. Abdou Zarzour, Halle
  - Universitätsklinikum Hamburg- Eppendorf, Institut für Versorgungsforschung in der Dermatologie und bei Pflegeberufen (IVDP), Hamburg
  - MVZ Prof. Dr. Ockenfels, Haut und Allergie-Praxisklinik GmbH, Hanau
  - Klinikum Region Hannover GmbH, KRH Klinikum Siloah, Klinik für Nephrologie, Angiologie und Rheumatologie, Hanover
  - Zentrum für Dermatochirurgie, St. Josefskrankenhaus Heidelberg GmbH, Heidelberg
  - SRH Klinikum Karlsbad- Langensteinbach GmbH, Interdisziplinäres Gefäßzentrum Innere Medizin, Karlsbad
  - Medizinisches Versorgungszentrum DermaKiel GmbH, Kiel
  - Hautarztpraxis Langenau, Studienzentrum, Langenau
  - Universitätsklinikum Leipzig AöR, Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Leipzig
  - Diabetologikum Ludwigshafen, die Praxis am Ludwigsplatz, Ludwigshafen
  - Beldio Research GmbH, Memmingen
  - Klinikum der Ludwig-Maximilians-Universität München, Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Universitätsklinikum Münster, Klinik für Hautkrankheiten, Allgemeine Dermatologie und Venerologie, Münster
  - Klinikum Nürnberg Nord, Klinik für Dermatologie, Nuremberg
  - MVZ Corius Potsdam GmbH, Dermatologie Potsdam MVZ, Potsdam
  - Caritas-Krankenhaus St. Josef, Klinik für Plastische und Ästhetische, Hand- und Wiederherstellungschirurgie, Regensburg
  - Universitätsmedizin Rostock, Klinik und Poliklinik für Dermatologie und Venerologie, Rostock
  - Helios Kliniken Schwerin, Plastische, Rekonstruktive und Ästhetische Chirurgie, Schwerin
  - Hautärztliche Gemeinschaftspraxis Dr. Leitz und Kollegen, Stuttgart
  - Universitätsklinikum Tübingen, Universitäts-Hautklinik Tübingen, Tübingen
  - Helios Universitätsklinikum Wuppertal, Zentrums für Dermatologie, Allergologie und Dermatochirurgie, Wuppertal
  - Universitätsklinikum Würzburg, Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Würzburg

IPD SHARING:
Plan to Share IPD: No